CLINICAL TRIAL: NCT04590755
Title: Run, Daddy, Run! A Multicomponent eHealth Lifestyle Intervention for the Prevention of Overweight and Obesity: Engaging Fathers and Their Children
Brief Title: Run Daddy Run! A Lifestyle Intervention Focusing on Fathers and Their Children
Acronym: RDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FWO17/ASP/123
Record Dates: First submitted 2020-09-09; First posted 2020-10-19 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-09

CONDITIONS: Father-Child Relations
Keywords: Obesity; Fathers; Children; Primary school; Intervention; Physical activity; Screen time; Sedentary Behaviour
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Non-Randomized Controlled Trial with Intervention and Control Group
Who Masked: Participant
Masking Description: Participants are allocated to the intervention or control group by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive father-child sessions and use of website (Experimental): Intervention group will receive the Run Daddy Run intervention.
  Interventions: Behavioral: Interactive father-child sessions and website
- No intervention (no interactive father-child sessions and use of website) (No Intervention): Intervention group will not receive the Run Daddy Run intervention.

INTERVENTIONS:
Behavioral: Interactive father-child sessions and website — The Run Daddy Run intervention will consist of 5 (inter)active sessions for fathers and their children + 1 follow-up session, each session lasting 90 minutes. These sessions will be given to 8 groups of +- 13 families (fathers and their children), guided by 2 facilitators and will take place every 2 weeks, at a location in the neighborhood of fathers and children (e.g. school of the children). Additionally, a website will be available for the fathers and their children, with additional information about the project, tips and information about being active together (e.g. movement breaks, fundamental movement skills, etc.) and limiting screen time. In addition, fathers and their children will also log their goals on this website, and between two sessions (= a period of 2 weeks) they will be asked to keep track of their co-PA on this website, aiming to reach their goal.
  Arms: Interactive father-child sessions and use of website

SUMMARY:
The aim of this study is to develop and implement a multicomponent eHealth lifestyle intervention (focusing on (co-) physical activity and screen time) for fathers and their children, aiming to prevent childhood overweight and obesity.

DETAILED DESCRIPTION:
The Run Daddy Run project aims to develop an effective lifestyle intervention for Belgian fathers and their primary school-aged children, to prevent overweight and obesity. There is focused on increasing (co-) physical activity and limiting individual and joint screen time. The project specifically targets fathers and their children because the literature shows that now often only mothers participate in lifestyle interventions, and fathers are underrepresented and difficult to involve. However, fathers play an important and unique role, independently of the mother, in shaping the child's behavior.

The Run Daddy Run intervention was developed based on the Intervention Mapping Protocol, a theoretical framework that is often used to develop interventions in a systematic way using empirical evidence and theoretical insights. A co-creation approach was also used for the intervention development, which is a bottom-up approach in which the target group (fathers in this case) is actively involved in the development of the intervention. The result of this approach is contextually appropriate intervention and intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Fathers
* Primary school aged children

Exclusion Criteria:

- Unhealthy/disease

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male: fathers Children: all (both boys and girls)
Enrollment: 102 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in co-physical Activity | 8 months (post-test), 14 months (follow-up)
  Father-child co-physical activity, will be subjectively measured using a seven-day recall diary, in which fathers will be asked to report all physical activities and screen time activities they performed together with their child in the last 7 days. More specifically, fathers have to report the start hour of the activity/activities, duration of the activity/activities, and the activity/activities itself in this diary, for each day of the week. PA diaries are often economical and can provide information on the types of activity not recorded from more objective measurement methods, such as accelerometers [66]. According to Matthews et al. (2002), diary based self-reported instruments can provide, with good participation compliance, accurate and valid assessments of PA [67].
Change in physical activity father | 8 months (post-test)
  Objective PA data will be collected through accelerometry. Axivity's (model AX3, 3-axial) will be worn by the father and the child for at least 7 consecutive days, on the non-dominant hand, for 24 hours a day. Participants' light (LPA), moderate (MPA), vigorous (VPA) and total PA will be assessed during this time period, which have been shown to be reliable and valid [60]. As an additional measure of (self-report) PA, fathers will be asked to complete the International Physical Activity Questionnaire Short Form (IPAQ-SF), for both himself and his child, questioning LPA, MPA and VPA during the past seven days [61, 62].Research comparing the IPAQ-SF with objective measures (i.e. accelerometers) shows that the criterion validity of this questionnaire is fair to good, with an ICC 0.30 [62]. Overall, the IPAQ-SF has reasonable (test-retest) reliability (ICC=0.65) a good internal consistency (Cronbach's Alpha=0.83) [63].
Change in physical activity child | 8 months (post-test)
  Objective PA data will be collected through accelerometry. Axivity's (model AX3, 3-axial) will be worn by the father and the child for at least 7 consecutive days, on the non-dominant hand, for 24 hours a day. Participants' light (LPA), moderate (MPA), vigorous (VPA) and total PA will be assessed during this time period, which have been shown to be reliable and valid [60]. As an additional measure of (self-report) PA, fathers will be asked to complete the International Physical Activity Questionnaire Short Form (IPAQ-SF), for both himself and his child, questioning LPA, MPA and VPA during the past seven days [61, 62].Research comparing the IPAQ-SF with objective measures (i.e. accelerometers) shows that the criterion validity of this questionnaire is fair to good, with an ICC 0.30 [62]. Overall, the IPAQ-SF has reasonable (test-retest) reliability (ICC=0.65) a good internal consistency (Cronbach's Alpha=0.83) [63].

SECONDARY OUTCOMES:
Change in co-screen time | 8 months (post-test)
  Co-ST will be measured using a seven-day recall diary, in which fathers will be asked to report all physical activities and screen time activities they performed together with their child in the last 7 days. More specifically, fathers have to report the start hour of the activity/activities, duration of the activity/activities, and the activity/activities itself in this diary, for each day of the week. PA diaries are often economical and can provide information on the types of activity not recorded from more objective measurement methods, such as accelerometers [66]. According to Matthews et al. (2002), diary based self-reported instruments can provide, with good participation compliance, accurate and valid assessments of PA [67].
Change in Sedentary behaviour (including screen time) father | 8 months (post-test)
  For measuring SB of the father, objective data will also be collected through accelerometry described under "Physical activity" measurements. Participants' SB will be assessed during a 7 days period using Axivity's, which have been shown to be a reliable and valid measure for SB. Additionally, SB (including ST) will be assessed using the International Sedentary Assessment Tool (ISAT) questionnaire [64]. This questionnaire has a good internal consistency (reliability) (Cronbach Alpha=0.80) and good criterion validity (interclass correlation r=0.63) [65]. In the ISAT, SB is questioned on week- and weekend days, as well as specific ST-related behaviours are questioned (i.e. TV/DVD viewing, computer/laptop/PlayStation use and smartphone/tablet use). The mean daily SB and ST of the fathers and their children will be calculated using the following formula: (SG or ST weekdays × 5 + SG or ST weekend days × 2) / 7.
Change in Sedentary behaviour (including screen time) child | 8 months (post-test)
  For measuring SB of the child, objective data will also be collected through accelerometry described under "Physical activity" measurements. Participants' SB will be assessed during a 7 days period using Axivity's, which have been shown to be a reliable and valid measure for SB. Additionally, SB (including ST) will be assessed using the International Sedentary Assessment Tool (ISAT) questionnaire [64]. This questionnaire has a good internal consistency (reliability) (Cronbach Alpha=0.80) and good criterion validity (interclass correlation r=0.63) [65]. In the ISAT, SB is questioned on week- and weekend days, as well as specific ST-related behaviours are questioned (i.e. TV/DVD viewing, computer/laptop/PlayStation use and smartphone/tablet use). The mean daily SB and ST of the fathers and their children will be calculated using the following formula: (SG or ST weekdays × 5 + SG or ST weekend days × 2) / 7.
Change in Father-child relationship (quality of relationship) | 8 months (post-test), 14 months (follow-up)
  Quality of the relationship between the father and the child will be measured with the Nurturant Fathering scale (NFS) [69]. This scale is a valid and reliable measure to characterize the relationship between the father and the child [70-72]. It consists of 9 items, each rated on a 5-point scale, and possible scores on this measure range from 9 to 45. Higher scores mean a better relationship.
Change in psychosocial determinants (co)PA | 8 months (post-test), 14 months (follow-up)
  The following determinants were questioned: (1) knowledge regarding the PA norm for both adults and (2) children, (3) knowledge and (4) self-efficacy towards motivating child for PA, (5) knowledge regarding limiting ST and (6) interrupting SB, (7) attitude towards limiting ST, (8) attitude towards and (9) importance of co-PA, (10) self-efficacy towards increasing co-PA, (11) degree of experienced barriers towards co-PA, (12) social support towards co-PA and (13) habits towards co-PA. For determinants on knowledge, participants were asked to estimate the norm (in minutes). The deviation from the norm was then calculated, with the value 0 representing a correct estimate of the norm and the higher the score deviating from 0, the greater the deviation from the correct answer. The other determinants were questioned and rated on a numerical response scale (values between 0 and 100, with 0 as the lowest score and 100 as the highest score).
Change in Family Health Climate | 8 months (post-test), 14 months (follow-up)
  The family context regarding PA will be questioned using the Family Health Climate Scale (FHC-PA) [68]. The family health climate can be seen as a determinant of person's health behaviour, and is defined as shared perceptions and cognitions concerning a healthy lifestyle within a family, and represents a family level variable that is intra- and inter-individually correlated to family environmental and individual factors. The FHC-PA is a validated questionnaire containing three subscales: value, cohesion and information on PA in the family. In total, this questionnaire contains 14 items, where participants can score these items on a 4-point Likert scale ranging from 1 "definitely false" to 4 "definitely true". The total score is the sum of all individual items scores, ranging from 14 to 56. Higher scores mean a better family health climate.
Change in Parental Practices regarding PA | 8 months (post-test), 14 months (follow-up)
  Parental skills and practices towards PA will be questioned in 16 questions, derived from four valid and reliable questionnaires each measuring specific parenting practices and skills [73-77].

CONTACTS AND LOCATIONS:
Overall Officials: Greet Cardon, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latomme J, Morgan PJ, Chastin S, Brondeel R, Cardon G. Effects of a family-based lifestyle intervention on co-physical activity and other health-related outcomes of fathers and their children: the 'Run Daddy Run' intervention. BMC Public Health. 2023 Feb 15;23(1):342. doi: 10.1186/s12889-023-15191-z. PMID 36793044
- [Derived] Latomme J, Morgan PJ, De Craemer M, Brondeel R, Verloigne M, Cardon G. A Family-Based Lifestyle Intervention Focusing on Fathers and Their Children Using Co-Creation: Study Protocol of the Run Daddy Run Intervention. Int J Environ Res Public Health. 2021 Feb 13;18(4):1830. doi: 10.3390/ijerph18041830. PMID 33668562